CLINICAL TRIAL: NCT02106585
Title: Phase 1, Randomized, Single-blind, Placebo-controlled Dose Escalation Study Evaluating Safety, Tolerability and Pharmacokinetics (PK) of JTT-251 Single Oral Doses in Healthy Subjects (Part Ia) and in Type 2 Diabetic Subjects (Part Ib) and Randomized, Open-label, Crossover Study Evaluating Effect of Food on PK in Healthy Subjects (Part II)
Brief Title: Study of Safety, Tolerability and Pharmacokinetics of Single Oral JTT-251 Doses in Healthy and Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT251-U-13-001
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus
Keywords: Safety; Tolerability; Pharmacokinetics; Food-effect; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (9):
- Dose 1 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 2 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 3 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 4 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 5 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 6 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 7 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 8 JTT-251 or Placebo (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-251 or Placebo
- Dose 9 JTT-251 or Placebo (Experimental): Tablets, single dose in fasted or fed condition followed by a single dose in the alternate fed or fasted condition
  Interventions: Drug: JTT-251 or Placebo

INTERVENTIONS:
Drug: JTT-251 or Placebo — Subjects will receive JTT-251 or Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK (Pharmacokinetics) of single oral doses of JTT-251 in healthy and type 2 diabetes mellitus subjects and to evaluate the effect of food on the PK of JTT-251 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subject Cohorts:

* Healthy male or female subjects
* Body Mass Index (BMI) between 19.0 and 31.0 kg/m2 (inclusive)

Type 2 Diabetic Subject Cohorts:

* Male or female Type 2 diabetic subjects diagnosed for at least 3 months
* BMI between 25 and 40 kg/m2 (inclusive)
* Have a glycosylated hemoglobin (HbA1c) of >6.5% to ≤10.9% (inclusive) if treatment naïve with respect to hypoglycemic agents OR >6.5% to ≤10.0% (inclusive) if treated with metformin

Exclusion Criteria:

Healthy Subject Cohorts:

* Known clinically relevant history or presence of significant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic, and dermatological or connective tissue disease
* Subjects with a systolic blood pressure >150 mmHg and/or diastolic blood pressure >90 mmHg

Type 2 Diabetic Subject Cohorts:

* Subjects with a known medical history or presence of type 1 diabetes mellitus
* Subjects with known medical history of acute metabolic diabetic complications
* Subjects with uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >95 mmHg with documented ongoing treatment)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 1 week
Vital signs and 12 lead ECGs | 1 week
Cmax (maximum concentration) | 1 week
t1/2 (elimination half-life) | 1 week
AUC (area under the concentration-time curve) | 1 week
fe(total) (fraction of systemically available drug excreted into the urine over entire collection interval) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Yamamoto, Study Chair — Akros Pharma Inc.
Locations (1):
- Orlando, Florida, United States